CLINICAL TRIAL: NCT04804605
Title: A Phase 3, Multicenter, Open-Label Extension Study of the Long-Term Safety of ARQ-151 Cream 0.15% and ARQ-151 Cream 0.05% in Subjects With Atopic Dermatitis
Brief Title: Open Label Extension Trial of PDE4 Inhibition With Roflumilast for the Management of Atopic Dermatitis
Acronym: INTEGUMENT-OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-313
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis Eczema
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-151 Cream 0.05% (Experimental): Participants applied ARQ-151 Cream 0.05% once daily (qd) for up to 52 weeks.
  Interventions: Drug: ARQ-151 Cream 0.15% or ARQ-151 Cream 0.05%

INTERVENTIONS:
Drug: ARQ-151 Cream 0.15% or ARQ-151 Cream 0.05% — ARQ-151 Cream 0.15% or ARQ-151 Cream 0.05%
  Other Names: Roflumilast

SUMMARY:
This study was a Phase 3, multicenter, open-label extension study of the long-term safety of roflumilast cream 0.15% (completers of studies ARQ-151-311 or ARQ-151-312 aged ≥6 years and ARQ-151-315 rollovers who turned 6 years of age on study) or roflumilast cream 0.05% (ARQ-151-315 rollovers aged 2 to 5 years). Participants with mild to moderate atopic dermatitis (AD) applied roflumilast cream once daily (qd) for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. For adult subjects: Participants legally competent to sign and give informed consent. For pediatric and adolescent subjects: Informed consent of parent(s) or legal guardian, and, if age appropriate, assent by the subjects, as required by local laws.
2. Males and females, ages 2 years and older. (Only subjects 18 years and older will be enrolled at sites located in the province of Québec in Canada.)
3. Subjects with atopic dermatitis who met eligibility criteria for and successfully completed one of three preceding studies through Week 4, and are able and eligible to enroll into this long-term safety study on the Week 4 visit of the preceding study.
4. Females of childbearing potential (FOCBP) must have a negative urine pregnancy test at all study visits. In addition, sexually active FOCBP must agree to use at least one form of a highly effective or barrier method of contraception throughout the trial.
5. Females of non-childbearing potential should either be pre-menarchal, or post-menopausal with spontaneous amenorrhea for at least 12 months (post-menopausal status would have been confirmed with FSH testing in the preceding study) or have undergone surgical sterilization (permanent sterilization methods include hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).
6. Subjects and parent(s)/legal guardian(s) are considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects who experienced a treatment-related AE or a serious AE (SAE) that precluded further treatment with ARQ-151 cream in the preceding study.
2. Subjects that use any Excluded Medications and Treatments.
3. Subjects with skin conditions other than AD that would interfere with evaluations of the effect of the study medication on AD, as determined by the Investigator. Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
4. Subjects with known genetic dermatological conditions that overlap with AD.
5. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
6. Subjects and parent(s)/legal guardian(s) who are unable to communicate, read or understand the local language(s), or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
7. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled subjects (subjects enrolled in other studies of ARQ-151 cream) living in the same house.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (92):
- United States (76):
  - Arcutis Clinical Site 112, Birmingham, Alabama
  - Arcutis Clinical Site 73, Birmingham, Alabama
  - Arcutis Clinical Site 63, Scottsdale, Arizona
  - Arcutis Clinical Site 106, Bryant, Arkansas
  - Arcutis Clinical Site 116, Fort Smith, Arkansas
  - Arcutis Clinical Site 69, Beverly Hills, California
  - Arcutis Clinical Site 81, Inglewood, California
  - Clinical Site 08, San Francisco, California
  - Arcutis Clinical Site 31, Santa Monica, California
  - Arcutis Clinical Site 130, Thousand Oaks, California
  - Arcutis Clinical Site 123, Centennial, Colorado
  - Arcutis Clinical Site 59, Coral Gables, Florida
  - Arcutis Clinical Site 72, Coral Gables, Florida
  - Arcutis Clinical Site 79, Delray Beach, Florida
  - Arcutis Clinical Site 103, Hollywood, Florida
  - Clinical Site 04, Jacksonville, Florida
  - Arcutis Clinical Site 15, Largo, Florida
  - Arcutis Clinical Site 67, Miami, Florida
  - Arcutis Clinical Site 95, Miami, Florida
  - Arcutis Clinical Site 68, Miami, Florida
  - Arcutis Clinical Site 29, Sanford, Florida
  - Clinical Site 01, Tampa, Florida
  - Arcutis Clinical Site 138, Wellington, Florida
  - Arcutis Clinical Site 47, Sandy Springs, Georgia
  - Arcutis Clinical Site 145, Boise, Idaho
  - Arcutis Clinical Site 13, Rolling Meadows, Illinois
  - Arcutis Clinical Site 93, Clarksville, Indiana
  - Clinical Site 22, Plainfield, Indiana
  - Arcutis Clinical Site 114, West Lafayette, Indiana
  - Clinical Site 03, Louisville, Kentucky
  - Arcutis Clinical Site 80, Covington, Louisiana
  - Arcutis Clinical Site 85, Lake Charles, Louisiana
  - Arcutis Clinical Site 24, Metairie, Louisiana
  - Arcutis Clinical Site 76, Rockville, Maryland
  - Arcutis Clinical Site 94, Bay City, Michigan
  - Arcutis Clinical Site 88, Clarkston, Michigan
  - Arcutis Clinical Site 58, Clinton Township, Michigan
  - Arcutis Clinical Site 66, Detroit, Michigan
  - Arcutis Clinical Site 132, Troy, Michigan
  - Clinical Site 10, New Brighton, Minnesota
  - Arcutis Clinical Site 102, Saint Joseph, Missouri
  - Arcutis Clinical Site 62, Reno, Nevada
  - Arcutis Clinical Site 71, East Windsor, New Jersey
  - Arcutis Clinical Site 96, Kew Gardens, New York
  - Arcutis Clinical Site 82, Rochester, New York
  - Arcutis Clinical Site 19, High Point, North Carolina
  - Arcutis Clinical Site 17, Gresham, Oregon
  - Arcutis Clinical Site 108, Portland, Oregon
  - Arcutis Clinical Site 16, Portland, Oregon
  - Arcutis Clinical Site 14, Portland, Oregon
  - Arcutis Clinical Site 53, Hershey, Pennsylvania
  - Arcutis Clinical Site 64, Newtown Square, Pennsylvania
  - Arcutis Clinical Site 25, Pittsburgh, Pennsylvania
  - Arcutis Clinical Site 101, Johnston, Rhode Island
  - Arcutis Clinical Site 77, Charleston, South Carolina
  - Arcutis Clinical Site 41, Charleston, South Carolina
  - Clinical Site 33, North Charleston, South Carolina
  - Arcutis Clinical Site 91, Summerville, South Carolina
  - Arcutis Clinical Site 60, Murfreesboro, Tennessee
  - Arcutis Clinical Site 34, Arlington, Texas
  - Clinical Site 23, Austin, Texas
  - Arcutis Clinical Site 84, Bellaire, Texas
  - Arcutis Clinical Site 21, College Station, Texas
  - Arcutis Clinical Site 126, Frisco, Texas
  - Arcutis Clinical Site 118, Grapevine, Texas
  - Arcutis Clinical Site 48, Houston, Texas
  - Arcutis Clinical Site 35, Houston, Texas
  - Arcutis Clinical Site 109, Katy, Texas
  - Clinical Site 20, San Antonio, Texas
  - Arcutis Clinical Site 49, San Antonio, Texas
  - Arcutis Clinical Site 74, Orem, Utah
  - Arcutis Clinical Site 36, West Jordan, Utah
  - Arcutis Clinical Site 51, Burke, Virginia
  - Arcutis Clinical Site 40, Norfolk, Virginia
  - Arcutis Clinical Site 12, Spokane, Washington
  - Arcutis Clinical Site 133, Kenosha, Wisconsin
- Canada (16):
  - Arcutis Clinical Site 70, Calgary, Alberta
  - Arcutis Clinical Site 27, Surrey, British Columbia
  - Arcutis Clinical Site 55, Winnipeg, Manitoba
  - Arcutis Clinical Site 50, Fredericton, New Brunswick
  - Arcutis Clinical Site 43, Ajax, Ontario
  - Arcutis Clinical Site 52, London, Ontario
  - Clinical Site 11, Markham, Ontario
  - Clinical Site 46, Mississauga, Ontario
  - Arcutis Clinical Site 46, Montréal, Ontario
  - Arcutis Clinical Site 61, Peterborough, Ontario
  - Arcutis Clinical Site 54, Toronto, Ontario
  - Arcutis Clinical Site 39, Waterloo, Ontario
  - Clinical Site 09, Windsor, Ontario
  - Arcutis Clinical Site 26, Drummondville, Quebec
  - Arcutis Clinical Site 45, Montreal, Quebec
  - Arcutis Clinical Site 56, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were rolled over upon completion of parent studies ARQ-151-311 (NCT04773587), ARQ-151-312 (NCT03638258), and ARQ-151-315 (NCT04845620). Rollovers from 311/312 were analyzed separately from 315 rollovers.
Pre-assignment Details: Participants with atopic dermatitis were enrolled at 153 sites in the United States (US), Canada, and Poland.
Groups:
- ARQ-151-311/312: RC/RC 0.15% Group: Participants who received roflumilast cream 0.15% in parent studies received roflumilast 0.15% cream qd for up to 52 weeks in the present study.
- ARQ-151-311/312: VC/RC 0.15% Group: Participants who received vehicle cream in the parent studies received roflumilast 0.15% cream qd for up to 52 weeks in the present study.
- ARQ-151-315: RC/RC 0.05% or 0.15% Group: Participants who received roflumilast cream 0.05% or 0.15% in the parent study received roflumilast 0.15% cream qd for up to 52 weeks in the present study. Participants received 0.05% until the first study visit after turning 6 years of age, and were then switched to 0.15%.
- ARQ-151-315: VC/RC 0.05% or 0.15% Group: Participants who received vehicle cream in the parent study received roflumilast 0.05% or 0.15% cream qd for up to 52 weeks in the present study. Participants received 0.05% until the first study visit after turning 6 years of age, and were then switched to 0.15%.
Period: Overall Study
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
Started | 439 | 219 | 382 | 180
Completed | 289 | 145 | 254 | 123
Not Completed | 150 | 74 | 128 | 57
Not completed — Withdrawal by Subject | 46 | 26 | 37 | 21
Not completed — Lost to Follow-up | 47 | 21 | 30 | 17
Not completed — Lack of Efficacy | 28 | 11 | 37 | 8
Not completed — Adverse Event | 10 | 10 | 10 | 7
Not completed — Non-compliance | 8 | 3 | 5 | 1
Not completed — Physician Decision | 3 | 0 | 5 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Miscellaneous | 7 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: One participant discontinued from the VC/RC Group prior to dosing.
Groups:
- Total: Total of all reporting groups
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group | Total
Number analyzed (Participants) | 439 | 218 | 382 | 180 | 1219
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (16.4) | 20.5 (17.9) | 3.4 (1.11) | 3.4 (1.17) | 12.2 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 122 | 185 | 91 | 642
  Male | 195 | 96 | 197 | 89 | 577
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 34 | 70 | 25 | 204
  Not Hispanic or Latino | 361 | 182 | 310 | 155 | 1008
  Unknown or Not Reported | 3 | 2 | 2 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 1 | 1 | 8
  Asian | 63 | 35 | 30 | 15 | 143
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 58 | 31 | 58 | 22 | 169
  White | 272 | 139 | 262 | 137 | 810
  More than one race | 20 | 7 | 25 | 3 | 55
  Unknown or Not Reported | 19 | 6 | 6 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Treatment-emergent Adverse Event (TEAE)
Description: The number of participants with ≥1 TEAE(s) is reported.
Time Frame: Up to 52 weeks
Population: All treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
Number analyzed (Participants) | 439 | 218 | 382 | 180
Participants | 151 | 90 | 189 | 91

2. Secondary Outcome: Validated Investigator Global Assessment-Atopic Dermatitis (vIGA-AD) Score of 0 or 1 at Each Assessment
Description: The vIGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported as score of 0 'clear' to 4 'severe' ), with lower scores indicating reduced symptom severity and vice versa. Multiple imputation was used to handle missing data up to Week 24 or 52 for 24- and 52-week cohorts.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
Number analyzed (Participants) | 439 | 219 | 382 | 180
percentage of participants
  Week 4 | 40.1 [35.61 to 44.83] | 35.7 [29.60 to 42.36] | 37.7 [32.98 to 42.77] | 40.8 [33.88 to 48.20]
  Week 12 | 42.2 [37.42 to 47.08] | 36.9 [30.55 to 43.68] | 40.0 [35.10 to 45.07] | 53.0 [45.62 to 60.25]
  Week 24 | 48.2 [43.25 to 53.18] | 46.3 [39.27 to 53.48] | 46.4 [41.25 to 51.54] | 54.3 [46.72 to 61.75]
  Week 36: number analyzed (Participants) | 243 | 117 | 377 | 176
  Week 36 | 45.5 [38.75 to 52.33] | 49.6 [39.36 to 59.82] | 42.5 [37.31 to 47.82] | 47.6 [39.94 to 55.45]
  Week 52: number analyzed (Participants) | 242 | 117 | 377 | 176
  Week 52 | 47.9 [40.82 to 55.07] | 45.0 [34.99 to 55.41] | 50.4 [44.86 to 55.99] | 56.9 [48.53 to 64.83]

3. Secondary Outcome: Percentage of Participants With vIGA-AD Success
Description: The percentage of participants with vIGA-AD "success" is presented. Success is defined as vIGA-AD value of 0 or 1 plus a 2-grade improvement from baseline. Multiple imputation was used to handle missing data up to Week 24 or 52 for 24- and 52-week cohorts.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
Number analyzed (Participants) | 439 | 219 | 382 | 180
percentage of participants
  Week 4 | 30.8 [26.65 to 35.33] | 7.8 [4.86 to 12.23] | 28.7 [24.38 to 33.48] | 11.1 [7.32 to 16.57]
  Week 12 | 33.7 [29.25 to 38.46] | 15.8 [11.46 to 21.48] | 29.5 [25.12 to 34.33] | 24.9 [19.01 to 31.93]
  Week 24 | 39.7 [35.02 to 44.67] | 21.6 [16.30 to 28.15] | 36.1 [31.31 to 41.13] | 24.1 [18.16 to 31.22]
  Week 36: number analyzed (Participants) | 243 | 117 | 377 | 176
  Week 36 | 37.4 [31.01 to 44.30] | 23.5 [15.60 to 33.77] | 34.4 [29.50 to 39.61] | 22.4 [16.45 to 29.70]
  Week 52: number analyzed (Participants) | 242 | 117 | 377 | 176
  Week 52 | 42.7 [35.78 to 50.01] | 24.2 [16.20 to 34.53] | 42.5 [37.11 to 48.15] | 28.5 [21.41 to 36.79]

4. Secondary Outcome: Change From Baseline in Worst Itch-Numeric Rating Scale (WI-NRS) Score Over Time in Participants ≥12 Years of Age in Parent Study
Description: Change from baseline in WI-NRS score is reported. WI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale is from '0 to 10' ("no itch" to "worst imaginable itch"), with lower scores indicating reduced symptom severity and vice versa.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All randomized participants who were ≥12 years of age at the start of the parent studies are included.
Measure: Mean (Standard Deviation); unit: WI-NRS Score Change
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
Number analyzed (Participants) | 256 | 139 | 0 | 0
WI-NRS Score Change
  Week 4: number analyzed (Participants) | 229 | 127 | 0 | 0
  Week 4 | -2.1 (2.80) | -0.3 (2.23) |  |
  Week 12: number analyzed (Participants) | 189 | 113 | 0 | 0
  Week 12 | -2.4 (3.06) | -0.2 (2.65) |  |
  Week 24: number analyzed (Participants) | 151 | 86 | 0 | 0
  Week 24 | -2.7 (2.85) | -0.8 (2.69) |  |
  Week 36: number analyzed (Participants) | 104 | 51 | 0 | 0
  Week 36 | -2.6 (2.81) | -0.3 (2.40) |  |
  Week 52: number analyzed (Participants) | 73 | 29 | 0 | 0
  Week 52 | -3.2 (2.85) | -1.2 (2.41) |  |

5. Secondary Outcome: Percent Change From Baseline in EASI Score
Description: EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90%-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (severe disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All randomized participants with data available are included.
Measure: Mean (Standard Deviation); unit: Percent change in EASI score
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
Number analyzed (Participants) | 439 | 219 | 382 | 180
Percent change in EASI score
  Week 4: number analyzed (Participants) | 417 | 208 | 382 | 180
  Week 4 | -63.23 (39.702) | -36.93 (63.272) | -59.51 (40.684) | -41.29 (53.042)
  Week 12: number analyzed (Participants) | 375 | 191 | 382 | 180
  Week 12 | -68.39 (34.195) | -17.95 (152.845) | -62.02 (49.438) | -16.11 (241.787)
  Week 24: number analyzed (Participants) | 325 | 159 | 382 | 180
  Week 24 | -72.81 (34.462) | -33.34 (116.997) | -71.04 (36.124) | -32.65 (16.532)
  Week 36: number analyzed (Participants) | 155 | 71 | 382 | 180
  Week 36 | -73.81 (31.300) | -39.20 (104.744) | -69.75 (40.467) | -39.39 (148.094)
  Week 52: number analyzed (Participants) | 145 | 63 | 382 | 180
  Week 52 | -74.57 (35.160) | -27.94 (137.809) | -77.78 (35.095) | -52.36 (74.751)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: All treated participants are included.
Arm/Group | ARQ-151-311/312: RC/RC 0.15% Group | ARQ-151-311/312: VC/RC 0.15% Group | ARQ-151-315: RC/RC 0.05% or 0.15% Group | ARQ-151-315: VC/RC 0.05% or 0.15% Group
All-Cause Mortality (participants affected / at risk) | 0/439 | 0/218 | 0/382 | 0/180
Serious Adverse Events (participants affected / at risk) | 5/439 | 3/218 | 12/382 | 3/180
Other Adverse Events (participants affected / at risk) | 18/439 | 12/218 | 82/382 | 40/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARQ-151-311/312: RC/RC 0.15% Group (N=439) | ARQ-151-311/312: VC/RC 0.15% Group (N=218) | ARQ-151-315: RC/RC 0.05% or 0.15% Group (N=382) | ARQ-151-315: VC/RC 0.05% or 0.15% Group (N=180)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0
Abscess jaw (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Application site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARQ-151-311/312: RC/RC 0.15% Group (N=439) | ARQ-151-311/312: VC/RC 0.15% Group (N=218) | ARQ-151-315: RC/RC 0.05% or 0.15% Group (N=382) | ARQ-151-315: VC/RC 0.05% or 0.15% Group (N=180)
COVID-19 (Infections and infestations) | 18 | 12 | 13 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 12 | 33 | 16
Nasopharyngitis (Infections and infestations) | 12 | 8 | 23 | 5
Pyrexia (General disorders) | 4 | 1 | 18 | 10
Influenza (Infections and infestations) | 7 | 3 | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The process of coordinating publication efforts is described in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT04804605/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT04804605/SAP_001.pdf